CLINICAL TRIAL: NCT02002806
Title: A Randomized Controlled Trial of Intraoperative Chemical Splanchnicectomy for Patients With Resected Pancreatobiliary Malignancies
Brief Title: Surgery Plus Celiac Nerve Block for Long-term Pancreatic Cancer Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Michael G. House, Associate Professor of Surgery, Indiana University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1011003552
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Pancreas Cancer; Biliary Tract Cancer
Keywords: Pancreatic cancer; Pain
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms; Pain | interventions — Ethanol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alcohol Injection (Experimental): Celiac plexus neurolysis by alcohol injection One time administration during surgery 20 ml of alcohol injection on each side of aorta at level of celiac axis
  Interventions: Other: Alcohol Injection
- Placebo Injection (Placebo Comparator): Celiac plexus injection - placebo injection
  Interventions: Other: Placebo Injection

INTERVENTIONS:
Other: Alcohol Injection — Celiac plexus neurolysis by alcohol injection
  Other Names: Ethanol Injection
  Arms: Alcohol Injection
Other: Placebo Injection
  Other Names: Normal saline injection
  Arms: Placebo Injection

SUMMARY:
This is a randomized study of surgery plus chemical nerve block versus surgery plus placebo for pain control in subjects with pancreatic cancer.

DETAILED DESCRIPTION:
Thi is a study of pain control in subjects undergoing surgery for pancreatic or bile duct cancer.

Subjects undergoing surgery will be randomized to surgery plus celiac plexus neurolysis with ethanol injection versus surgery plus placebo injection. Subjects will be followed every three months for survivorship or death to assess pain, quality of life measures, and narcotic pain control usage. The primary endpoint of pain control will be determined at one year post surgery. Subjects are not required to undergo any additional diagnostic testing procedures that are not part of their routine follow-up care.

ELIGIBILITY:
Inclusion Criteria:

This study will be offered to all patients scheduled to undergo open or laparoscopic operative resection of a presumed pancreatic (any location; i.e., head, body, or tail) or distal biliary tract cancer.

* Physiologic suitability for major abdominal surgery
* Aged 18 years and older
* Written informed consent
* Ability to understand and comply with study guidelines.

Exclusion Criteria:

* Pregnancy
* Previous, preoperative celiac nerve block
* Neoadjuvant chemotherapy or radiation therapy
* Incomplete tumor resection (R2 resection, grossly positive resection margin)
* Presumed ampullary or duodenal cancer based on preoperative work-up or intraoperative findings
* Benign tumors, neuroendocrine tumors, soft tissue tumors based on preoperative work-up or intraoperative findings
* Known metastatic disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-01; Primary Completion 2018-12 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Pain Control | 12 Months

SECONDARY OUTCOMES:
Disease-specific, recurrence-free survival | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Michael G House, MD, Principal Investigator — Indiana University, Department of Surgery
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No